CLINICAL TRIAL: NCT04885244
Title: Prospective Evaluation of Complex Adult Spinal Deformity (CAD) Treated With Minimally Invasive Surgery (MIS)
Brief Title: Prospective Evaluation of Complex Adult Spinal Deformity (CAD) Treated With Minimally Invasive Surgery
Acronym: MIS
Status: Recruiting | Type: Observational
Sponsor: International Spine Study Group Foundation (Other)
Collaborators: NuVasive (Industry)
Responsible Party: Sponsor
Other Study IDs: 2138
Record Dates: First submitted 2021-05-10; First posted 2021-05-13 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Adult Spinal Deformity; Scoliosis; Kyphosis; Sagittal Imbalance
Keywords: Scoliosis; Kyphosis; Sagittal Imbalance; Spinal Deformity
MeSH Terms: conditions — Scoliosis; Kyphosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Operative: Multicenter, prospective, nonrandomized analysis of ASD patients w/diagnosis of congenital, degenerative, idiopathic, neuromuscular, inflammatory or iatrogenic spinal deformity. Participants must be scheduled to have 3 or more levels of Percutaneous posterior spinal instrumentation or 3 level stand alone lateral surgery within next 6 months.
  Interventions: Procedure: Index or spine revision surgery for complex adult spinal deformity

INTERVENTIONS:
Procedure: Index or spine revision surgery for complex adult spinal deformity — Surgical interventions will be patient specified by treating surgeon.

SUMMARY:
Evaluate surgical treatment outcomes and identify best practice guidelines for complex adult spinal deformity (ASD) patients treated with minimally invasive approach, including radiographic and clinical outcomes, surgical and postoperative complications, risk factors for and revision surgery rates, and the role of standard work to improve patient outcomes and reduce surgical and postoperative complications.

DETAILED DESCRIPTION:
Specific Aims:

* Evaluate surgical treatment outcomes and identify best practice guidelines for complex adult spinal deformity (ASD) patients treated with minimally invasive approach, including radiographic and clinical outcomes, surgical and postoperative complications, risk factors for and revision surgery rates, and the role of standard work to improve patient outcomes and reduce surgical and postoperative complications.

  a. Complex ASD patients will be defined based upon clinical, radiographic and/or procedural criteria.
* Develop and validate a standardized, universal complications classification system for minimally invasive spine surgery
* Evaluate perioperative blood management approaches, transfusion requirements, including variance in thresholds for blood transfusion and associated complications for minimally invasive adult spinal deformity surgery
* Evaluate clinical outcomes utilizing legacy patient reported outcome measures (PROMs) including Scoliosis Research Society 22r (SRS 22r) modified Oswestry Disability Index (mODI), Veterans RAND-12 (VR-12), and numeric pain rating scale (NRS), and patient reported outcome measurement information system (PROMIS).
* Evaluate clinical outcomes stratifying by patient chronological and physiological age
* Evaluate the cost for episode of care for minimally invasive CADS surgery and cost per QALY gain compared to open surgery for CADS
* Evaluate the contribution of patient frailty to patient outcomes, cost of care, disability, and complications
* Evaluate incidence of and risk factors for mental health (MH) compromise among ASD patients treated with MIS techniques, and establish best practice guidelines for assessing MH
* Evaluate the association of MH with surgical complications, outcomes, hospital length of stay and cost for MIS ASD surgery
* Evaluate the association of social health surgical complications, outcomes, hospital length of stay and cost for MIS ASD surgery and risk factors for routine (home) discharge vs. skilled nursing facility (SNF)/rehabilitation facility
* Broaden the evaluation of the minimally invasive surgically treated ASD patient to maximize evaluation of the entirety of the episode of care to include steps that can be taken prior to surgery including "prehabilitation," pain management, and MH care to improve treatment outcomes, reduce cost, reduce hospital length of stay, reduce non-routing discharge and reduce early and late complications
* Establish a core set of standard work guidelines to clinically and radiographically evaluate and treat ASD patients and evaluate the utility of standard work to improve outcomes for ASD and formulate best practice guidelines for minimally invasive surgical treatment of ASD
* Evaluate the use of robotic techniques in minimally invasive spine surgery for ASD, and its impact on radiographic parameters and clinical outcomes
* Evaluate the use of expandable cages in minimally invasive spine surgery for ASD, and its impact on radiographic parameters and clinical outcomes
* Evaluate the OR efficiency, morbidity of surgery, and cost per episode of care relating to single-position vs. multi-position CADS surgery
* Evaluate the prevalence and incidence of sacroiliac pain before/after complex adult spinal deformity surgery.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years of age at the time of treatment 2. Diagnosis of adult congenital, degenerative, idiopathic, neuromuscular, inflammatory or iatrogenic spinal deformity 3. EOS full body or standing 36" AP & Lateral images of entire spine 4. Surgery to be schedule to take place within 6 months (otherwise PROMs/Radiographic images to be recollected) 5. Surgery to include > 3 levels percutaneous posterior spinal instrumentation or 3 level stand-alone lateral 6. And any one of the following:

a. Radiographic criteria incorporating percutaneous posterior spinal instrumentation: i. PI-LL ≥ 25 degrees ii. Thoracolumbar/lumbar scoliosis ≥ 20 degrees iii. SVA >10cm iv. PT > 30 b. Procedural criteria: i. Single-position surgery ≥ 3 levels fused (Levels=vertebra; S1 is counted as a level; S2 &/or pelvis/ilium is not) ii. Staged ≥ 3 levels fused with percutaneous pedicle screws iii. 3 column osteotomy with percutaneous fixation iv. ACR incorporating open or percutaneous fixation

Exclusion Criteria:

1. Deformity due to acute trauma
2. Active spine tumor or infection
3. Patient is unwilling or unable to complete questionnaires
4. Women who are pregnant
5. Prisoners -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multi-center, prospective, non-randomized analysis of surgically treated complex adult spinal deformity (ASD) patients
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-07-28 (Actual); Primary Completion 2034-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Scoliosis Research Society (SRS) 22r | Change from Preop to 3 months and 1, 2, 5 & 10 year follow-up
  Scoliosis specific patient reported outcome
Oswestry Disability Index (ODI) | Change from Preop to 3 months and 1, 2, 5 & 10 year follow-up
  Spine specific patient reported outcome
Veterans RAND 12 Item Health Survey (VR-12) | Change from Preop to 3 months and 1, 2, 5 & 10 year follow-up
  Patient reported outcome
Patient-Reported Outcome Measurement Information System (PROMIS) - Anxiety | Change from Preop to 3 months and 1, 2, 5 & 10 year follow-up
  Computer adaptive Patient reported outcome
Patient-Reported Outcome Measurement Information System (PROMIS) - Depression | Change from Preop to 3 months and 1, 2, 5 & 10 year follow-up
  Computer adaptive Patient reported outcome
Patient-Reported Outcome Measurement Information System (PROMIS) - Pain Interference | Change from Preop to 3 months and 1, 2, 5 & 10 year follow-up
  Computer adaptive Patient reported outcome
Patient-Reported Outcome Measurement Information System (PROMIS) - Physical Function | Change from Preop to 3 months and 1, 2, 5 & 10 year follow-up
  Computer adaptive Patient reported outcome
Patient-Reported Outcome Measurement Information System (PROMIS) - Social Satisfaction | Change from Preop to 3 months and 1, 2, 5 & 10 year follow-up
  Computer adaptive Patient reported outcome
Patient-Reported Outcome Measurement Information System (PROMIS) - Social Role Satisfaction | Change from Preop to 3 months and 1, 2, 5 & 10 year follow-up
  Computer adaptive Patient reported outcome
Radiographic Evaluation | Change from Preop to 3 months and 1, 2, 5 & 10 year follow-up
  Cobb angles, Coronal & Sagittal balance, spinopelvic measures
Visual Analog Scale - Back Pain | Change from Preop to 3 months and 1, 2, 5 & 10 year follow-up
  Self-reported back pain on scale of 0 (No pain) to 10 (severe pain)
Visual Analog Scale - Leg pain | Change from Preop to 3 months and 1, 2, 5 & 10 year follow-up
  Self-reported leg pain on scale of 0 (No pain) to 10 (severe pain)

SECONDARY OUTCOMES:
Edmonton Frail Scale | Change from Preop to 3 months and 1, 2, 5 & 10 year follow-up]
  Evaluate frailty on scale of 0 to 17 where higher scores mean more frail
Canadian Study of Health and Aging (CSHA) | Change from Preop to 3 months and 1, 2, 5 & 10 year follow-up]
  Frailty scale of 1 to 9; higher scores mean more frail
Adverse Events | Change from Preop to 3 months and 1, 2, 5 & 10 year follow-up]
  Occurrence of Adverse events meeting reporting criteria and their relationship to intervention throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Praveen Mummaneni, MD, Principal Investigator — University of San Francisco; Paul Park, MD, Principal Investigator — University of Michigan; Gregory Mundis, MD, Principal Investigator — Scripps Clinic, Department of Orthopedic Surgery, La Jolla, CA; Juan Uribe, MD, Principal Investigator — Barrow Neurological Institute, Phoenix, AZ
Locations (12):
- United States (12):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Shiley Center for Orthopaedic Research and Education at Scripps Clinic, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California - San Francisco Medical Center, San Francisco, California
  - University of Miami, Miami, Florida
  - Rush University, Department of Neurosurgery, Chicago, Illinois
  - Louisiana Spine Institute, Shreveport, Louisiana
  - University of Michigan, Department of Neurosurgery, Ann Arbor, Michigan
  - Columbia University - New York-Presbyterian Och Spine Hospital, New York, New York
  - Duke University Health System, Durham, North Carolina
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Semmes-Murphey, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No